CLINICAL TRIAL: NCT02615366
Title: Minimization of Bleeding Complications Through Utilization of Perioperative Tranexamic Acid in Breast Surgery: A Randomized Double-blinded Placebo-controlled Trial
Brief Title: Tranexamic Acid for Bleeding in Breast Surgery
Acronym: TABBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20150264-01H
Record Dates: First submitted 2015-11-17; First posted 2015-11-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Hematoma; Seroma
MeSH Terms: conditions — Hematoma; Seroma | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): Tranexamic acid will be provided as an intravenous infusion (1g in 100mL 0.9% NaCl solution [1% TXA] at 5 ml/min) 20 minutes pre-operatively, followed by an additional intravenous dose of the same dosing parameters postoperatively. Oral tablet doses containing 1 g of TXA (2x 500mg tablets) per dose will be administered to the patient to be taken orally by the patient according to a standard regimen; the first tablet dose will be taken on the same day as the surgery, in the evening. The patient will then take one tablet dose three times a day for a total of five days following the surgery (one dose in the morning, one dose mid-day, and one dose in the afternoon) for a 6 day total regimen.
  Interventions: Drug: Tranexamic Acid
- Placebo Control (Placebo Comparator): Placebo control will be either 100 ml of 0.9% NaCl solution or tablets of similar appearance containing no medicinal ingredients; placebo will be administered according to the same regimen as the intervention group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo
  Arms: Placebo Control

SUMMARY:
Bleeding is an important consideration in breast surgeries that involve large resections of soft tissues in the breast. Inappropriate bleeding during or after surgery, can lead to uncomfortable fluid buildup in the breasts known as a hematoma or seroma, which may require additional procedures or reoperation. Patients may experience a great deal of discomfort and additional costs as a result; additional hospital time and procedures also burdens health care spending. Tranexamic acid (TXA) is commonly used drug in many medical settings to reduce excessive bleeding; however, no such drug is standard practice in breast surgery. The aim of this study is to determine if TXA is superior to placebo in reducing the bleeding complications in breast surgeries, including reduction mammaplasty, mastectomy with and without immediate tissue expander and implant-based reconstruction, and oncoplastic breast surgery. This study is a randomized, double-blind, placebo-controlled trial. Patients undergoing these procedures will be randomly allocated to receive either TXA or placebo. Patients will be placed on a drug/placebo regimen of 3 doses/day for 6 days starting on the day of their surgery. The primary outcome is the incidence of hematoma and/or seroma formation following breast surgery. Cost analysis of the intervention will also be performed.

DETAILED DESCRIPTION:
Background:

Aberrant bleeding is an important consideration in breast surgery, which can involve large resections of soft tissues in the breasts. Hematomas and/or seromas are common complications with these procedures, and can lead to further complications, such as flap necrosis. Seromas, perhaps the commonest complication, are documented to occur at rates as high as 85% in certain breast procedures. Hematoma rates are typically lower than that of seroma, ranging from 1% to 2% in mastectomy procedures and 5% to 8% in reduction mammaplasty. These bleeding complications pose an obvious risk to patient safety, and their management can result in significant costs to patients and healthcare alike.

Tranexamic acid (TXA), also known by the brand name Cyklokapron® from Pfizer™, is a lysine analogue used to prevent and/or treat bleeding by competitively blocking the activation of plasminogen to plasmin, thereby preventing plasmin from binding to blood clots. Tranexamic acid is used safely in several medical and surgical settings, such as cone biopsies, epistaxis and hyphaema control, and dental surgery. This antifibrinolytic medication is commonly used in many surgical procedures, namely cardiac and orthopedic surgery, for the purposes of preventing blood loss. TXA has been demonstrated to effectively reduce perioperative blood loss and transfusion rates in many different surgical procedures, such as cardiac, urology, gynecology, and orthopedic surgeries, without any significant safety concerns.

Despite these findings, there is a clear paucity of studies on TXA in breast surgery. There are currently no studies exploring perioperative TXA use in breast reduction, and only one study in breast surgery overall. This study by Oertli et al. looked at the use of TXA in mastectomy or lumpectomy with axial dissection, in a randomized placebo-controlled trial (RCT). Seroma rate was shown to be reduced by 10% with a reduction in TXA versus placebo. However, due to a low power of the study, Oertli et al. were unable to determine statistical significance.

Purpose:

The purpose of this study is to determine if perioperative administration of tranexamic acid (TXA) is superior to placebo in minimizing bleeding complications (as determined by: hematoma/seroma incidence in the breast, re-operation and/or additional procedures, blood transfusion volume, drainage volume (Jackson-Pratt drain or percutaneous drainage), number of days spent in hospital) in breast surgery (Reduction mammaplasty, mastectomy with and without immediate tissue expander and implant-based reconstruction, oncoplastic breast surgery). Conterminous with this objective, the investigators also intend to study the safety of tranexamic acid use perioperatively in these procedures by recording any adverse effects that occur at the time of surgery and throughout the follow-up period. The study will randomize and prospectively observe two patient populations undergoing any one of these procedures: one group receiving preoperative and subsequent post-operative 1g doses of tranexamic acid, and the other receiving placebo (normal saline). These two groups will be observed based on specific properties and complications from surgery. Finally, to determine if perioperative TXA use is more cost-effective than placebo in the setting of breast surgery. Information on health care utilization will be collected prospectively in both groups to provide a cost analysis of tranexamic acid.

The following hypotheses will be tested:

1. Perioperative TXA use is superior to placebo in reducing bleeding complications (ie. hematoma, seroma, and excessive blood loss) in the surgical or donor site.
2. Perioperative TXA is safe for use in this patient population.

Study Design

The present study will be a randomized, double-blind, placebo-controlled trial. This RCT will follow the CONSORT statement. Conterminous to this RCT, data on treatment costs (hospital and patient cost) will be recorded. The study will last approximately two years. Case Report Forms will be filled out at each follow-up period. Follow-up will occur at 2 weeks, 6 weeks, and 12 weeks postoperatively. Cost-analysis of the intervention will also be performed.

Sample Size:

Based on published data, the incidence of the combined hematoma/seroma endpoint is expected to range between 6 and 10% in the reductions patients and 16-87% in the mastectomy patients. Since the investigators expect to have equal numbers of each type of patient, the investigators anticipate the overall event rate in the placebo arm to range between 11-47%. Taking the midpoint, the investigators anticipate a placebo arm event rate of 29%. The investigators would consider a 30% relative reduction (i.e., an absolute difference of 9%) to be the minimal clinically important difference that would, if demonstrated, change practice. To detect this difference with 80% power, the investigators require 385 patients per arm using a two-sided test at the 5% level of significance To account for attrition of 15 patients per arm (<5%), the investigators will aim to 400 patients per group.

Data Analysis:

The unit of analysis will be each individual patient for all outcomes. Baseline characteristics will be compared between study arms using descriptive statistics (frequencies and proportions for categorical variables, mean and standard deviation for continuous variables with a normal distribution and median and inter-quartile range for variables with a skewed distribution). The investigators' primary outcome, the incidence of hematoma and/or seroma, will be analyzed using a chi-square test with continuity correction. The difference between the arms will be described using a relative risk with 95% confidence interval. The overall rate in each group will also be reported. Secondary outcomes will be analyzed using chi-square tests (dichotomous outcomes) or Wilcoxon tests (drainage volume, transfusion volume, and days in hospital). Drainage and transfusion volume, as well as the number of days in hospital, will be summarized as median and interquartile range. All data analysis will be carried out by a statistician from the Ottawa Hospital Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires and is a candidate for any of the following surgical procedures: Reduction mammaplasty, mastectomy with and without immediate tissue expander and implant-based reconstruction, oncoplastic breast surgery.
* Patient has OHIP approval for surgery.
* Patient is willing and able (ie. English/French-speaking and cognitively intact) to read and complete patient diaries, demographic forms, and consent forms and be followed-up for a 2 weeks, 6 weeks, 12 weeks postoperatively.
* Patient is 18 years of age or older

Exclusion Criteria:

* Patient is allergic to tranexamic acid
* Patient has a history or present laboratory signs of bleeding disorders (abnormal platelet counts, prothrombin time, partial thromboplastin time, etc.), coagulopathy or thromboembolic events
* Patient is being treated for a stroke
* Patient has a history of bleeding in the brain
* Patient has an acquired disturbance of colour vision
* Patient has a history of myocardial infarction within the last year
* Patient is presenting with unstable angina or severe coronary disease
* Patient has reduced renal function with plasma creatinine levels above 250 umol/L ix.
* Patient has haematuria
* Patient is currently using a form of birth control that contains estrogen and a progestin
* Patient has irregular menstrual bleeding of unknown cause
* Patient is unable to complete required forms due to language and cognitive problems
* Patient is not capable of communicating in, and understanding, English or French
* Patient is currently pregnant and is expected to be pregnant during any point of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of hematoma or seroma formation in breast surgical site as assessed by clinical examination. | 12 weeks following the operation
  Hematoma or seroma formation in the breast surgical site(s) will be identified by surgeon on clinical examination during patient follow-up within 12 weeks post-operatively.

SECONDARY OUTCOMES:
Tranexamic Acid Adverse Events: | 12 weeks following the operation
  Includes allergic and/or anaphylactic reactions, eye or eyesight problems, thromboembolic events, diarrhoea, gastrointestinal problems, hypersensitivity reactions, nausea and vomiting
Drainage volume as measured from Jackson-Pratt drain or percutaneous drainage | 12 weeks following the operation
Blood transfusion volume | During surgical operating time, during post-operative hospital admission time (1-7 days on average).
Incidence of secondary breast operation | 12 weeks following the operation
  Surgical revision of initial breast procedure due to unsatisfactory results
Incidence of additional procedures following initial breast operation to address hematoma or seroma | 12 weeks following the operation
  Operative or non-operative procedures to correct hematoma or seroma in the breast surgical site
Number of days spent in hospital | 12 weeks following the operation
Cost associated with bleeding complications | 12 weeks following the operation
  Additional cost of original procedure (including material costs, as well as OR time, surgeon, anesthetist, and nurse costs), cost per day spent in hospital, cost for additional care (including procedures, medication, etc.), patient/caregiver out-of-pocket expenses (dressings and medications, parking, transportation, days missed from work)

REFERENCES:
- [Background] Taylor JC, Rai S, Hoar F, Brown H, Vishwanath L. Breast cancer surgery without suction drainage: the impact of adopting a 'no drains' policy on symptomatic seroma formation rates. Eur J Surg Oncol. 2013 Apr;39(4):334-8. doi: 10.1016/j.ejso.2012.12.022. Epub 2013 Feb 4. PMID 23380200
- [Background] de la Pena-Salcedo JA, Soto-Miranda MA, Lopez-Salguero JF. Prophylactic mastectomy: is it worth it? Aesthetic Plast Surg. 2012 Feb;36(1):140-8. doi: 10.1007/s00266-011-9769-x. Epub 2011 Jul 13. PMID 21751064
- [Background] Lovely JK, Nehring SA, Boughey JC, Degnim AC, Donthi R, Harmsen WS, Jakub JW. Balancing venous thromboembolism and hematoma after breast surgery. Ann Surg Oncol. 2012 Oct;19(10):3230-5. doi: 10.1245/s10434-012-2524-y. Epub 2012 Jul 21. PMID 22820939
- [Background] Alani HA, Balalaa N. Complete tissue expander coverage by musculo-fascial flaps in immediate breast mound reconstruction after mastectomy. J Plast Surg Hand Surg. 2013 Oct;47(5):399-404. doi: 10.3109/2000656X.2013.772060. Epub 2013 Jun 26. PMID 23802185
- [Background] Lapid O, Pietersen L, van der Horst CM. Reoperation for haematoma after breast reduction with preoperative administration of low-molecular-weight heparin: experience in 720 patients. J Plast Reconstr Aesthet Surg. 2012 Nov;65(11):1513-7. doi: 10.1016/j.bjps.2012.05.027. Epub 2012 Jun 23. PMID 22728066
- [Background] Pannucci CJ, Wachtman CF, Dreszer G, Bailey SH, Portschy PR, Hamill JB, Hume KM, Hoxworth RE, Kalliainen LK, Rubin JP, Pusic AL, Wilkins EG. The effect of postoperative enoxaparin on risk for reoperative hematoma. Plast Reconstr Surg. 2012 Jan;129(1):160-168. doi: 10.1097/PRS.0b013e318236215c. PMID 21915085
- [Background] Carpelan A, Kauhanen S, Mattila K, Jahkola T, Tukiainen E. Reduction mammaplasty as an outpatient procedure: a retrospective analysis of outcome and success rate. Scand J Surg. 2015 Jun;104(2):96-102. doi: 10.1177/1457496914526872. Epub 2014 May 7. PMID 24809356
- [Background] Xu Q, Yang Y, Shi P, Zhou J, Dai W, Yao Z, Zhang C. Repeated doses of intravenous tranexamic acid are effective and safe at reducing perioperative blood loss in total knee arthroplasty. Biosci Trends. 2014 Jun;8(3):169-75. doi: 10.5582/bst.2014.01063. PMID 25030852
- [Background] Gillette BP, DeSimone LJ, Trousdale RT, Pagnano MW, Sierra RJ. Low risk of thromboembolic complications with tranexamic acid after primary total hip and knee arthroplasty. Clin Orthop Relat Res. 2013 Jan;471(1):150-4. doi: 10.1007/s11999-012-2488-z. PMID 22814857
- [Background] Oertli D, Laffer U, Haberthuer F, Kreuter U, Harder F. Perioperative and postoperative tranexamic acid reduces the local wound complication rate after surgery for breast cancer. Br J Surg. 1994 Jun;81(6):856-9. doi: 10.1002/bjs.1800810621. PMID 8044602
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893